CLINICAL TRIAL: NCT05100810
Title: A Monocentric, Prospective, Longitudinal and Observational Natural History Study for Patients With Angelman Syndrome in the United Kingdom: Natural History - Foundation for Angelman Syndrome Therapeutics (FAST) United Kingdom (UK)
Brief Title: Angelman Syndrome Natural History Study-FAST UK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Foundation for Angelman Syndrome Therapeutics UK (Unknown); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: PID15397
Record Dates: First submitted 2021-08-13; First posted 2021-10-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Angelman Syndrome
Keywords: Natural History; EEG; ActiMyo; outcome measures; proteomics
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15 mls of blood will be collected during each visit. Blood samples will be centrifuged and plasma stored in the Department of Paediatrics, University of Oxford. Proteomics will be performed on plasma samples. Some blood will be collected for the Angelman Syndrome DNA biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Angelman syndrome patients: This study will comprehensively evaluate the natural clinical progression of the disease using scales and questionnaires for the assessment of motor function and global development, movement monitoring devices (ActiMyo), and by collecting sleep and seizure diaries. In addition, proteomic analysis and electroencephalography (EEG) recordings will be collected to identify biomarkers that will indicate improvements in disease outcome following treatment.
  Interventions: Other: Natural History Study

INTERVENTIONS:
Other: Natural History Study — Longitudinal assessment of disease progression of Angelman syndrome in patients

SUMMARY:
The goal of this study is to conduct a prospective, longitudinal assessment of the natural clinical progression of Angelman syndrome (AS) in children and adults. This will be performed by acquiring baseline measurements, and developing effective outcome measures and diagnostic tools for the syndrome, to prepare the healthcare system for forthcoming clinical trials.

DETAILED DESCRIPTION:
This study is being conducted in anticipation of several candidate therapies which are approaching clinical readiness for Angelman syndrome. This study will comprehensively evaluate the natural clinical progression of the disease using scales and questionnaires for the assessment of motor function and global development, motor measuring devices (ActiMyo), and by collecting sleep and seizure diaries. In addition, proteomic analysis and electroencephalography (EEG) recordings will be collected to identify biomarkers which will indicate improvements in disease outcome following treatment.

ELIGIBILITY:
Inclusion Criteria:

For the candidate participants affected by AS:

* Genetically confirmed diagnosis of AS
* 0-99 years
* Male or Female
* Obtained consent forms and/or record of consultation by the carers.

In this study, the two primary carers for each participant diagnosed with AS will be also considered participants. Carers will have to meet the following inclusion criteria:

* Male or Female
* >18 years
* Legal carer of the patient diagnosed with AS
* Willingness to follow study procedures, as assessed by the research team
* Willingness to sign the consent form
* Ability to understand all the information regarding the study, as assessed by the research team

Exclusion Criteria:

* The participant affected by AS may not enter the study if there is any comorbidity (*) that could potentially affect the results of the study. This will be subject to the clinical judgement of the Chief Investigator (CI) and/or the Principal Investigator (PI). Participants of ongoing (interventional) clinical trials that assess the efficacy of potential treatments will be excluded as assessments need to be done on the basis that represent the natural progression of AS.

(*) This includes any confirmed chronic or acute condition or disease affecting any system(s), which could interfere with the results of the study and/or the compliance with the study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Genetically confirmed diagnosis of AS
  * 0-99 years
  * Male or Female
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of relevant medical data (retrospective and prospective) | 2 years 1 month
  Collection of demographic data, Angelman Syndrome-related medical history, past medical and surgical history, current medication, history of immunisations and family medical history.
Neurological assessment scale | 2 years 1 month
  Hammersmith Infant Neurological Examination (HINE) (0-2 years ONLY). Maximum global score of 78. Higher scores indicate a higher degree of neurological performance.
Clinical Scale | 2 years 1 month
  Clinical Global Impressions Scale - Angelman Syndrome version (CGI-SAS). Scales whereby practitioner rates from 1 to 7 the overall improvement/deterioration of the participant affected by Angelman Syndrome. One is improved and 7 denotes deterioration.
Clinical Scale | 2 years 1 month
  Caregiver-reported Angelman Syndrome Scale (CASS). Scales whereby the carer rates from 1 to 7 the overall improvement/deterioration of the participant affected to by Angelman Syndrome. One is improved and 7 denotes deterioration.

SECONDARY OUTCOMES:
Movement monitoring using wearable device | 2 years 1 month
  Continuous movement monitoring using actimetry ActiMyo® in uncontrolled environment (i.e., home)
Gross motor milestones | 2 years 1 month
  World Health Organisation (WHO) Motor Milestones. Scale of 6 gross motor milestones. Lower scores denotes worse motor function.
Global development assessment scale | 2 years 1 month
  Bayley Scales of Infant and Toddler Development - 4 (BSID-4) for Developmental delays. Scale is divided into five domains, which are further divided into subdomains. The first step is to calculate the starting point by beginning with the items that are age appropriate. The starting point is validated if three consecutive items are achieved. If the participant affected by Angelman Syndrome does not achieve three consecutive items in a row at the age-appropriated starting point, the evaluator must go backwards to the lower age-starting point until the participant affected by Angelman Syndrome achieves three items in a row. The assessment stops once five items in a row are not achieved.
Global development assessment scale | 2 years 1 month
  Vineland Adaptive Behaviour Scales-III (VABS-III). Scale composed of two main domains, which are subdivided into several subdomains. Lower score indicates worse cognitive functioning.
Aberrant behaviour assessment | 2 years 1 month
  Aberrant Behaviour Checklist-Community (ABC-C). This scale comprises 58 items and is divided into five subdomains. The ABC-C is designed on a four-point scale with the lowest score representing less-affected patients while the highest score represents the severest patients.
Communication assessment | 2 years 1 month
  Observed Reported Communication Assessment (ORCA) Tool. Questionnaire designed to be completed by the patients' main carer and records patient communication.
Motor function assessment | 2 years 1 month
  Functional Mobility Scale (FMS). Scale which rates the walking ability in three different walking distances, and these distances will be rated on a 6-point scale.
Sleep and seizure activity | 2 years 1 month
  Sleep and seizure diaries with ready-made questionnaires
Laboratory biomarkers for Angelman syndrome | 2 years 1 month
  Proteomic analysis of plasma samples to determine biomarkers of disease progression
Electroencephalogram (EEG) activity recordings | 24 hours
  Electroencephalogram (EEG) to record brain activity of Angelman Syndrome patients over a 24-hour period (e.g., sleep architecture, number and frequency of seizures, background epileptic activity, delta-rhythmicity)
Quality of Life questionnaires for families of Angelman syndrome patients | 2 years 1 month
  PedsQL-Family Module questionnaires. Questionnaire uses ranking system of 1-4 based on frequency.
Quality of life assessment for individuals affected by Angelman syndrome | 2 years 1 month
  PedsQL-Core Module questionnaires. Questionnaire uses ranking system which depends on the age of patient.
Health economics | 2 years and 1 month
  Interview with Carer's
Clinical trial readiness | 2 years and 1 month
  Demographic data collection and facilities preparation

OTHER OUTCOMES:
DNA biobank | 2 years and 1 month
  Blood sample collection and DNA extraction and storage

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, OXON, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided